CLINICAL TRIAL: NCT02122549
Title: Hospital Wearable Defibrillator Inpatient Study
Acronym: HWD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 90D0118
Record Dates: First submitted 2014-04-17; First posted 2014-04-24 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-02

CONDITIONS: In-Hospital Cardiac Arrest
Keywords: In-Hospital Cardiac Arrest; Telemetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HWD1000 (Experimental): Subjects using HWD1000
  Interventions: Device: HWD1000

INTERVENTIONS:
Device: HWD1000 — Wearable cardioverter-defibrillator designed for inpatient use

SUMMARY:
This study will obtain device-human interaction evaluations for the HWD1000 within the controlled environment of the hospital as well as establish that the safety profile is similar to outpatient wearable cardioverter-defibrillators use.

DETAILED DESCRIPTION:
A multi-center prospective study of hospitalized patients whom a physician deems at risk of sudden cardiac arrest during the hospitalization period, wearing the HWD1000 hospital wearable defibrillator in order to evaluate caregiver and patient interactions with the device. In addition, ECG signal quality will be reviewed to confirm the HWD1000 safety profile.

ELIGIBILITY:
Inclusion Criteria:

Patients whom a physician deems at risk of sudden cardiac arrest during the hospitalization period (patients will be monitored using the hospital's telemetry system). Specific inclusion criteria are:

* Hospitalized patients having continuous independent ECG monitoring.
* Patients at risk of sudden cardiac arrest during the hospitalization period as determined by the investigating physician.
* Patient ≥18 years of age (over the legal age of providing consent).

Exclusion Criteria:

* Patients with an active implantable cardioverter-defibrillator.
* Patients with an active unipolar pacemaker.
* Patients with physical or mental conditions preventing them from interacting with or wearing the device as determined by the investigating physician.
* Patients having an advanced directive prohibiting resuscitation.
* Patients having bandages or other clinical condition preventing the HWD use.
* Patients unable to consent.
* Patients having recently experienced an arrhythmic storm.
* Patients prone to paroxysmal supraventricular tachycardia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Szymkiewicz, MD, Principal Investigator — Zoll Medical Corporation
Locations (8):
- United States (8):
  - Los Angeles, California
  - Danbury, Connecticut
  - Atlantis, Florida
  - Jupiter, Florida
  - Iowa City, Iowa
  - Saint Paul, Minnesota
  - Richmond, Virginia
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HWD1000
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Hospitalized patients at risk for sudden cardiac arrest.
Arm/Group | HWD1000
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Rhythm Monitoring by the HWD1000 is Compromised Due to ECG Noise.
Description: The amount of time that the HWD1000 is unable to monitor the subject's rhythm status is the primary safety measure. The specific goals are that average monitoring will be inhibited by noise no greater than 2% of the time worn (at least 24 hours) and monitoring using single lead analysis will be no greater than 5% of the time worn (at least 24 hours).
Time Frame: 24 hours or longer
Population: Subjects who wore the HWD 1000 for a minimum of 24 hours.
Measure: Mean (Standard Deviation); unit: percentage of time worn
Groups:
- HWD1000: Subjects wearing the HWD 1000.
Arm/Group | HWD1000
Number analyzed (Participants) | 38
percentage of time worn
  Neither lead used for monitoring | 0.53 (0.73)
  One lead not used for monitoring | 2.54 (3.16)

ADVERSE EVENTS:
Arm/Group | HWD1000
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HWD1000 (N=59)
Skin Iritation (Skin and subcutaneous tissue disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days